CLINICAL TRIAL: NCT03097211
Title: A Double-blind, Randomised, Placebo-controlled, Rising Multiple Dose Study in Healthy Volunteers to Investigate the Effect of BIA 6-512 at Steady-state on the Levodopa Pharmacokinetics When Administered in Combination With a Single-dose of Levodopa/Benserazide 200/50 mg or With a Single-dose of Levodopa/Benserazide 200/50 mg Plus a Single-dose of Nebicapone 150 mg
Brief Title: Effect of BIA 6-512 at Steady-state on the Levodopa Pharmacokinetics With a Single-dose of Levodopa/Benserazide 200/50 mg or With a Single-dose of Levodopa/Benserazide 200/50 mg Plus a Single-dose of Nebicapone 150 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-6512-107
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Resveratrol; benserazide, levodopa drug combination; nebicapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: BIA 6-512 25 mg or placebo (Experimental): Subjects were administered with those investigational products at approximately 8-h intervals, starting in the morning (approximately at 8h00) of Day 1 and finishing in the morning of Day 5 (last dose). On Day 4, concomitantly with the BIA 6-512/Placebo morning dose, one tablet of Madopar® 250 was administered. On Day 5, concomitantly with the BIA 6-512/Placebo morning dose, one tablet of Madopar® 250 and one tablet of nebicapone 150 mg were administered
  Interventions: Drug: Placebo; Drug: BIA 6-512; Drug: Madopar® 250; Drug: Nebicapone
- Group 2: BIA 6-512 50 mg or placebo (Experimental): Subjects were administered with those investigational products at approximately 8-h intervals, starting in the morning (approximately at 8h00) of Day 1 and finishing in the morning of Day 5 (last dose). On Day 4, concomitantly with the BIA 6-512/Placebo morning dose, one tablet of Madopar® 250 was administered. On Day 5, concomitantly with the BIA 6-512/Placebo morning dose, one tablet of Madopar® 250 and one tablet of nebicapone 150 mg were administered
  Interventions: Drug: Placebo; Drug: BIA 6-512; Drug: Madopar® 250; Drug: Nebicapone
- Group 3: BIA 6-512 75 mg or placebo (Experimental): Subjects were administered with those investigational products at approximately 8-h intervals, starting in the morning (approximately at 8h00) of Day 1 and finishing in the morning of Day 5 (last dose). On Day 4, concomitantly with the BIA 6-512/Placebo morning dose, one tablet of Madopar® 250 was administered. On Day 5, concomitantly with the BIA 6-512/Placebo morning dose, one tablet of Madopar® 250 and one tablet of nebicapone 150 mg were administered
  Interventions: Drug: Placebo; Drug: BIA 6-512; Drug: Madopar® 250; Drug: Nebicapone
- Group 4: BIA 6-512 100 mg or placebo (Experimental): Subjects were administered with those investigational products at approximately 8-h intervals, starting in the morning (approximately at 8h00) of Day 1 and finishing in the morning of Day 5 (last dose). On Day 4, concomitantly with the BIA 6-512/Placebo morning dose, one tablet of Madopar® 250 was administered. On Day 5, concomitantly with the BIA 6-512/Placebo morning dose, one tablet of Madopar® 250 and one tablet of nebicapone 150 mg were administered
  Interventions: Drug: Placebo; Drug: BIA 6-512; Drug: Madopar® 250; Drug: Nebicapone

INTERVENTIONS:
Drug: Placebo — Placebo capsules. Orally, with 240 mL of potable water.
Drug: BIA 6-512 — The investigational products consisted of capsules containing BIA 6-512 25 mg, 50 mg, 75 mg, 100 mg. Orally, with 240 mL of potable water.
  Other Names: Trans-resveratrol
Drug: Madopar® 250 — Levodopa/benserazide immediate release tablets 200mg/50mg. Orally, with 240 mL of potable water.
  Other Names: Levodopa/benserazide
Drug: Nebicapone — Nebicapone 150 mg tablets. Orally, with 240 mL of potable water.
  Other Names: BIA 3-202

SUMMARY:
The purpose of this study was to determine whether the administration of BIA 6-512 (25 mg, 50 mg, 75 mg and 100 mg) at steady-state affects the pharmacokinetics of levodopa when administered in combination with a single-dose of immediate release levodopa/benserazide 200/50 mg or with a single-dose of immediate release levodopa/benserazide 200/50 mg plus a single-dose of nebicapone 150 mg.

DETAILED DESCRIPTION:
Single centre, double-blind, randomised, placebo-controlled, rising multiple dose study in four sequential groups of healthy male and female subjects. Eligible subjects were admitted to the Human Pharmacology Unit (UFH)on the day prior to receiving the first study medication. Starting in the morning of Day 1 (first dose), subjects received BIA 6-512/Placebo thrice daily until the morning of Day 5 (last dose). Concomitantly with the morning dose of BIA 6-512/Placebo on Day 4, a levodopa/benserazide 200/50 mg (Madopar® 250) single-dose was administered. On Day 5, a Madopar® 250 single-dose and a nebicapone 150 mg single-dose were administered concomitantly with the morning dose of BIA 6-512/Placebo. In the morning of Day 4 and Day 5, products were administered in fasting conditions of at least 8 hours and subjects remained fasted until 2 h post-dose. Subjects were resident in the UFH from admission (Day 0) until at least 24 h post last dose (Day 6); then, they were discharged and returned for the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Subjects who had negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening
* Subjects who had clinical laboratory test results clinically acceptable at screening and admission.
* Subjects who had a negative screen for alcohol and drugs of abuse at screening and admission.
* Subjects who were non-smokers or who smoked ≤ 10 cigarettes or equivalent per day.
* Subjects who were able and willing to gave written informed consent.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier, intrauterine device or abstinence.
* (If female) She had a negative urine pregnancy test at screening and admission.

Exclusion Criteria:

* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 14 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening or admission.
* Subjects who had acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission.
* Subjects who had used medicines within 2 weeks of admission that may affect the safety or other study assessments, in the investigator's opinion.
* Subjects who had previously participated in a clinical trial with BIA 6-512.
* Subjects who had used any investigational drug or participated in any clinical trial within 6 months prior to screening.
* Subjects who had participated in more than 2 clinical trials within the 12 months prior to screening.
* Subjects who had donated or received any blood or blood products within the 3 months prior to screening.
* Subjects who were vegetarians, vegans or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not use an effective contraceptive method (double-barrier, intra-uterine device or abstinence) or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2006-07-17 (Actual); Primary Completion 2006-10-20 (Actual); Study Completion 2006-10-20

PRIMARY OUTCOMES:
Day 4 - Maximum observed plasma drug concentration (Cmax) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8 and 16 hours post-dose.
  Pharmacokinetic parameters of BIA 6-512, levodopa, and nebicapone on day 4
Day 4 - Time of occurrence of Cmax (tmax) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8 and 16 hours post-dose.
  Pharmacokinetic parameters of BIA 6-512, levodopa, and nebicapone on day 4
Day 4 - Area under the plasma concentration-time curve (AUC) from time zero to the last sampling time at which concentrations were at or above the limit of quantification (AUC0-t) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8 and 16 hours post-dose.
  Pharmacokinetic parameters of BIA 6-512, levodopa, and nebicapone on day 4
Day 4 - AUC from time zero to 8 h post-dose (AUC0-τ) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8 and 16 hours post-dose.
  Pharmacokinetic parameters of BIA 6-512, levodopa, and nebicapone on day 4
Day 4 - Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8 and 16 hours post-dose.
  Pharmacokinetic parameters of BIA 6-512, levodopa, and nebicapone on day 4
Day 4 - Apparent terminal elimination half-life, calculated from ln 2/λz (t1/2) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8 and 16 hours post-dose.
  Pharmacokinetic parameters of BIA 6-512, levodopa, and nebicapone on day 4
Day 5 - Maximum observed plasma drug concentration (Cmax) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 16 and 24 hours post-dose
  Pharmacokinetic parameters of BIA 6-512, levodopa, and nebicapone on day 5
Day 5 - Time of occurrence of Cmax (tmax) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 16 and 24 hours post-dose
  Pharmacokinetic parameters of BIA 6-512, levodopa, and nebicapone on day 5
Day 5 - Area under the plasma concentration-time curve (AUC) from time zero to the last sampling time at which concentrations were at or above the limit of quantification (AUC0-t) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 16 and 24 hours post-dose
  Pharmacokinetic parameters of BIA 6-512, levodopa, and nebicapone on day 5
Day 5 - AUC from time zero to 8 h post-dose (AUC0-τ) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 16 and 24 hours post-dose
  Pharmacokinetic parameters of BIA 6-512, levodopa, and nebicapone on day 5
Day 5 - Area under the plasma concentration versus time curve from time zero to infinity (AUC0-∞) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 16 and 24 hours post-dose
  Pharmacokinetic parameters of BIA 6-512, levodopa, and nebicapone on day 5
Day 5 - Apparent terminal elimination half-life, calculated from ln 2/λz (t1/2) | pre-dose, ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 16 and 24 hours post-dose
  Pharmacokinetic parameters of BIA 6-512, levodopa, and nebicapone on day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Human Pharmacology Unit (UFH) - BIAL - Portela & Cª, SA, S. Mamede Do Coronado, Portugal

IPD SHARING:
Plan to Share IPD: Undecided